CLINICAL TRIAL: NCT00310141
Title: Treatment of Nicotine Dependence Among African Americans
Brief Title: Computer-Assisted Counseling in Helping African American Smokers Stop Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ID01-234; R01CA094826 (NIH); P30CA016672 (NIH); MDA-ID-01234 (Other: UT MD Anderson Cancer Center); CDR0000466339 (Registry Identifier: NCI PDQ); NCI-2012-01637 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Counseling; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Care Group (Active Comparator): Written self-help materials, counseling, and 6-week nicotine patch supply
  Interventions: Other: Counseling intervention; Drug: Nicotine patch
- Computer Treatment Group (CDT) (Active Comparator): Written self-help materials, counseling, 6-week nicotine patch supply and 6 weeks of computer-delivered treatment
  Interventions: Behavioral: Smoking cessation intervention; Other: Counseling intervention; Drug: Nicotine patch
- CDT Pilot (Experimental): Written self-help materials, counseling, 6-week nicotine patch supply and 6 weeks of computer-delivered treatment
  Interventions: Behavioral: Smoking cessation intervention; Other: Counseling intervention; Drug: Nicotine patch

INTERVENTIONS:
Behavioral: Smoking cessation intervention — 6 weeks of computer delivered treatment for quitting smoking
  Arms: CDT Pilot; Computer Treatment Group (CDT)
Other: Counseling intervention — In-person counseling (5 sessions)
Drug: Nicotine patch — 6-week supply of the nicotine patch

SUMMARY:
RATIONALE: Stop-smoking plans using a nicotine patch, in-person counseling, and computer-assisted counseling may help people stop smoking.

PURPOSE: This randomized clinical trial is studying how well computer-assisted counseling helps African American smokers stop smoking.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop and evaluate the efficacy of an interactive, culturally sensitive, individualized, palmtop computer-delivered smoking cessation intervention for African American smokers.
* Examine how hypothesized treatment mechanisms mediate the effects of computer-delivered treatment on abstinence.

OUTLINE: This is a randomized study. A subset of 20 participants are assigned to arm II for pilot testing. All other participants are randomized to 1 of 2 intervention arms.

* Arm I (standard care [SC]): Participants receive nicotine patch therapy on days -5 to 31. Participants also receive a Pathways to Freedom self-help guide and undergo 5 in-person counseling sessions based on the Treating Tobacco Use and Dependence Clinical Practice Guideline. The counseling sessions occur at 12 and 5 days prior to the quit smoking date and at 3, 10, and 31 days after the quit smoking date.
* Arm II (computer-delivered treatment [CDT]): Participants receive the same intervention as in arm I. Participants also undergo CDT for 6 weeks comprising 5 modules (quitting strategies; motivation and support; general smoking information; calendars and fun stuff; and daily tips) beginning 12 days prior to the quit smoking date and continuing for 31 days after the quit smoking date.

All participants complete questionnaires at baseline, during the counseling sessions, and then at approximately 6 months after the quit smoking date.

After completion of study intervention, participants are followed at approximately 6 months.

PROJECTED ACCRUAL: A total of 500 participants will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. African American
2. Age 21 to 65 years
3. Current Smoker (history of at least 5 cigarettes/day for the last year)
4. Motivated to quit within the next 14 days
5. Participants must provide a viable home address and functioning home telephone number
6. Can speak, read, write in English at a sixth-grade literacy level
7. Provide viable collateral contact information
8. Register "8" or more on a carbon monoxide breath test

Exclusion Criteria:

1. Contraindication for nicotine patch use
2. Active substance dependence (exclusive of nicotine dependence)
3. Regular use of tobacco products other than cigarettes (cigars, pipes, smokeless)
4. Use of bupropion or nicotine products other than nicotine patches supplied by the study
5. Pregnancy or lactation
6. Any active illness that precludes full participation in the study protocol
7. Another household member enrolled in the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2002-04-08 (Actual); Primary Completion 2006-08-17 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Smoking status by SRNT Smoking Status Questionnaire 6 months after treatment | 6 months after treatment
  Abstinence measures are collected at four post cessation follow-up visits. Point prevalence serving as the primary outcome measure. Primary outcome analyses will use data from all of the follow-up visits. SRNT Abstinence Status Questionnaire (Hughes et al., 2003) surveys the tobacco use by the participant and persons within the participant's household and social surroundings. The questionnaire also collects data on the use of other tobacco products and nicotine replacement medications. The pre- and post-quit versions of this questionnaire have been adapted to specific timepoints corresponding to participant visits.

SECONDARY OUTCOMES:
Contemplating smoking by Contemplation Ladder 6 months after treatment | 6 months after treatment
  The Contemplation Ladder (Biener & Abrams, 1991) assesses readiness to quit smoking and ranges from 0-10 with 0 being "no thought of quitting" and 10 being "taking action to quit" (e.g., cutting down, enrolling in a program).

CONTACTS AND LOCATIONS:
Overall Officials: David W. Wetter, PhD, MS, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org